CLINICAL TRIAL: NCT04428957
Title: Telemonitoring as a Tool for the Assessment of Treatment Effects of Connective Tissue Disease-associated Interstitial Lung Disease (TEL-CTD-ILD)
Brief Title: Telemonitoring of Treatment Effects in Connective Tissue Disease-associated Interstitial Lung Disease (TEL-CTD-ILD)
Acronym: TEL-CTD-ILD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RNN/50/20/KE; 0047/DW/2018 (Other Grant/Funding Number: Polish Ministry of Science and Higher Education)
Record Dates: First submitted 2020-04-08; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-04

CONDITIONS: Connective Tissue Disease-associated Interstitial Lung Disease; Interstitial Lung Disease; Connective Tissue Diseases
Keywords: Telemonitoring; Telemedicine; Interstitial lung disease; Connective Tissue Diseases; Treatment
MeSH Terms: conditions — Lung Diseases, Interstitial; Connective Tissue Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemonitoring group (Experimental): 3 months home-based telemonitoring
  Interventions: Other: Telemonitoring
- Control group (No Intervention): 3 months standard care

INTERVENTIONS:
Other: Telemonitoring — Daily telemonitoring of heart rate (HR), blood pressure (BP), pulse oximetry (SpO2), spirometry (FVC), activity (accelerometry) and severity of cough and dyspnea
  Arms: Telemonitoring group

SUMMARY:
1. Impact of telemonitoring on quality of life (QoL) of patients with CTD-ILD
2. Evaluation of health status of patients with connective tissue disease-associated interstitial lung disease (CTD-ILD) using telemonitoring and standard care.
3. Assessment of treatment response patterns (full remission, partial remission, progression, no response) and evaluation of clinical prognostic factors (risk factors for poor response in patients with CTD-ILD.
4. Evaluation of cost-effectiveness of telemonitoring solutions in patients with CTD-ILD.
5. Evaluation of telemedicine as a tool for assessing the safety of therapy

DETAILED DESCRIPTION:
Interstitial lung disease (ILD) is one of the most serious pulmonary complications related to connective tissue diseases (CTDs), resulting in substantial morbidity and mortality. Interstitial lung disease is a common manifestation of different connective tissue diseases, such as scleroderma, rheumatoid arthritis (RA), Sjögren's syndrome, systemic lupus, dermatomyositis and others. Radiological and histopathological patterns are most often nonspecific interstitial pneumonia (NSIP), organizing pneumonia (OP), usual interstitial pneumonia (UIP) and lymphocytic interstitial pneumonia (LIP).

Current standard of care in progressive CTD associated ILD is low to medium dose of corticosteroids, frequently combined with immunosuppressive medication, depending on disease severity and local standards. However, based on clinical and radiological features, it is difficult to predict what will be the response to the treatment. Effectiveness of the treatment is assessed by functional tests and chest high resolution computed tomography (HRCT), performed usually after 3 months of therapy.

Project objective is to assess the possible benefits of using telemonitoring of functional and vital signs, symptoms and quality of life of patients with CTD-ILD in response to treatment.

In the trial patients diagnosed with CTD-ILD will be randomized to intervention group (telemonitoring) and the control group (traditional assessment). Patients from the study after initial training will perform daily spirometry (FVC), transdermal pulse oximetry, pulse and blood pressure measurements, activity measurement (accelerometry), and assessment of severity of cough and dyspnea. The additional questionnaires will also be used to assess the tolerability of treatment, quality of life and the occurrence of side effects. Telemonitoring will start 10 to 14 days before the start of treatment and will be carried out for 3 months of therapy. All patients (study and control group) will receive treatment in accordance with current treatment standards. During the 3-month observation period, visits to the center will take place at monthly intervals. In the case of treatment intolerance or deterioration of monitored parameters, patients will be evaluated at additional time points. All patients after the end of the 3-month follow-up will remain under the care of the Pulmonology Clinic and will be examined during regular visits every 3 months until the end of the 12-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed interstitial lung disease with a small component of fibrous changes;
* Indications for systemic glucocorticoid therapy +/- immunosuppressant;
* 18 years and older
* Informed consent to participate in the study;
* Effective contraception;
* Result of the Mini Mental test ensuring the possibility of efficient operation of monitoring devices;
* Completed training in the operation of telemedicine equipment.

Exclusion Criteria:

* Evidence of irreversible interstitial fibrotic changes in lung HRCT;
* Pattern of definite or probable usual interstitial pneumonia (UIP) in the HRCT examination;
* Contraindications to glucocorticoid and immunosuppressive therapy (azathioprine or mycophenolate mofetil or cyclophosphamide or cyclosporine);
* Pregnancy and breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-02-11 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline health-related quality of life using EQ-5D-5L questionnaire at 3 months | at baseline, after 3 months
  The EuroQoL Group 5-Dimension 5-Level Self Report Questionnaire (EQ-5D-5L) questionnaire will be used for the assessment of quality of life. The EQ-5D-5L essentially consists of 2 pages - the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-5L is especially suited to cost effectiveness analyses.
Change from baseline health-related quality of life using St. George's Respiratory Questionnaire at 3 months | at baseline, after 3 months
  St. George's Respiratory Questionnaire (SGRQ) will be used to assess health related quality-of-life. The SGRQ is a 50-item questionnaire developed to measure health status (quality of life) in patients with diseases of airways obstruction. SGRQ is survey with scores ranging from 0 to 100 and with higher scores indicating worse quality of life.

SECONDARY OUTCOMES:
Costs of health service utilization in Polish zloty | after 3 months, after 6 months
  Mean costs in telemonitoring and control group will be estimated. Healthcare utilization will be assessed through the number of emergency department, hospital or outpatient clinic visits, medications and adverse events treatments. Resource use categories will be monetarily valued using unit cost and multiplied with the collected amount of resource use. Mean costs in Polish zloty per group will be calculated.
Assessment of Dyspnea using Modified Medical Research Council (mMRC) | at baseline, after 3 months
  The Modified Medical Research Council Dyspnea (mMRC) scale will be used to determine functional impairment due to dyspnea. It is a five-level rating scale consisting of just five items containing statements about the impact of dyspnea on the patients' daily activities performance. Higher scores indicate a greater impact of dyspnea on the patients' daily activities performance.
Assessment of fatigue using Fatigue Assessment Scale (FAS) | at baseline, after 3 months
  Fatigue Assessment Scale (FAS) will be used for assessment of fatigue status. The total score ranges from 10 to 50. A total FAS score < 22 indicates no fatigue, a score ≥ 22 indicates fatigue.
Assessment of patients' adherence to recommended medications using the Adherence Scale in Chronic Diseases (ASCD) | at baseline, after 3 months
  The Adherence Scale in Chronic Diseases is a self-reported questionnaire with 8 items and with proposed 5 sets of answers. The total score in the Adherence Scale in Chronic Diseases ranges from 0 to 32 points. Three levels of adherence were considered (low: scores of 0 to 20; medium 21 to 25; high > 26).
Change from baseline anxiety and depression symptoms as measured by HADS (Hospital Anxiety and Depression Scale) | at baseline, after 3 months
  The Hospital Depression and Anxiety Index (HADS) is a 14-item survey with scores ranging from 0 to 21 and with higher scores indicating greater depression and anxiety.
Change from baseline depression as measured by PHQ-9 | at baseline, after 3 months
  The Patient Health Questionnaire (PHQ-9) is a 10-item survey with scores ranging from 1 to 27 and with higher scores indicating greater levels of depression.
For the telemonitoring arm, oxygen saturation (SpO2) expressed in percent | twice a day day from baseline for 3 months
  Oxygen saturation level (SpO2) will be measured by transdermal Pulse Oximeter.
For the telemonitoring arm, heart rate (HR) expressed in beats per minute (bpm) | twice a day day from baseline for 3 months
  Heart rate home telemonitoring consisted of twice-daily patient self-measurement of heart rate with automated device.
For the telemonitoring arm, systolic blood pressure (SBP) expressed in mmHg | twice a day day from baseline for 3 months
  Systolic BP will be assessed by home-based blood pressure telemonitoring using sphygmomanometer
For the telemonitoring arm, diastolic blood pressure (DBP) expressed in mmHg | twice a day day from baseline for 3 months
  Diastolic BP will be assessed by home-based blood pressure telemonitoring using sphygmomanometer
For the telemonitoring arm, forced vital capacity (FVC) expressed in percent | twice a day day from baseline for 3 months
  Lung function like forced vital capacity (FVC, %FVC) will be assessed using home spirometry.
For the telemonitoring arm, forced expiratory volume in 1st second (FEV1) expressed in percent | twice a day day from baseline for 3 months
  Lung function like forced expiratory volume in 1 second (FEV1, ％FEV1) will be assessed using home spirometry.
For the telemonitoring arm, patient's satisfaction assessed by developed telemonitoring satisfaction survey. | after 3 months
  Developed telemonitoring satisfaction survey will be used for the assessment of patient's satisfaction in 10 areas assessed using the 5-point Likert scale.
For the telemonitoring arm, cough severity measured using 5-point Likert scale (range 0-4) | twice a day day from baseline for 3 months
  A 5-point Likert scale will be used to measure cough severity
For the telemonitoring arm, dyspnea severity measured using a 5-point Likert scale (range 0-4) | twice a day day from baseline for 3 months
  A 5-point Likert scale will be used to measure dyspnea severity

CONTACTS AND LOCATIONS:
Overall Officials: Wojciech Piotrowski, Assoc. Prof., Principal Investigator — Department of Pneumology and Allergy, Medical University of Lodz
Locations (1):
- Department of Pneumology and Allergy, Medical University of Lodz, Lodz, Lodz Province, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Malysiak-Szpond S, Mozga M, Miadlikowska E, Milkowska-Dymanowska J, Bialas AJ, Piotrowski WJ. Study protocol for connective tissue disease-associated interstitial lung disease trial (TEL-CTD-ILD): A randomized controlled trial of a home-based telemonitoring of treatment effects. PLoS One. 2022 Dec 27;17(12):e0278601. doi: 10.1371/journal.pone.0278601. eCollection 2022. PMID 36574413